CLINICAL TRIAL: NCT02142855
Title: Structural and Metabolic Determinants of Sarcopenia and the Efficacy of Concentric vs. Eccentric Exercise Training: a Novel Temporospatial Approach
Brief Title: Structural and Metabolic Determinants of Sarcopenia and the Efficacy of Concentric vs. Eccentric Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B13032014 SoMSGEM BBSRC3
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: volunteers; young (18-30 y); older (65-75 y); age groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Old Control (No Intervention): Older individuals (65-75 y) with no exercise intervention
- Old Concentric (Experimental): Older individuals (65-75 y) studied before and after 8 weeks concentric exercise training
  Interventions: Behavioral: Concentric Exercise Training
- Old Eccentric (Experimental): Older individuals (65-75 y) studied before and after 8 weeks eccentric exercise training
  Interventions: Behavioral: Eccentric Exercise Training
- Young Control (No Intervention): Young individuals (18-30 y) with no exercise intervention
- Young Concentric (Experimental): Young individuals (18-30 y) studied before and after 8 weeks concentric exercise training
  Interventions: Behavioral: Concentric Exercise Training
- Young Eccentric (Experimental): Young individuals (18-30 y) studied before and after 8 weeks eccentric exercise training
  Interventions: Behavioral: Eccentric Exercise Training

INTERVENTIONS:
Behavioral: Concentric Exercise Training — 8 weeks concentric exercise training, 3 x per week, 60% 1-RM; 4 x 12-15 repetitions, 2 min rest between sets
  Arms: Old Concentric; Young Concentric
Behavioral: Eccentric Exercise Training — 8 weeks eccentric exercise training, 3 x per week, 60% 1-RM; 4 x 12-15 repetitions, 2 min rest between sets
  Arms: Old Eccentric; Young Eccentric

SUMMARY:
The first goal of this study is the follow young and older people over a period of 8 weeks to define the processes responsible for loss of muscle length and width in age-related muscle wasting (sarcopenia) and allow us to look at age-related differences in tendon. Secondly, we will assess two different exercise interventions for reversing human sarcopenia; one which involves shortening of the muscle and the other which involves lengthening, whilst also studying why these exercises work the way they do. This project will have significant implications for our understanding of the control of skeletal muscle and tendon size in humans, particularly in relation to sarcopenia and the surrounding health issues.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Body mass index 18-30 kg/m2
* Aged 18-35 and 65-75 years

Exclusion Criteria:

* Participation in a formal exercise regime,
* A BMI < 18 or > 30 kg/m2,
* Active cardiovascular disease,
* Taking beta-adrenergic blocking agents, statins or non-steroidal anti-inflammatory drugs,
* Cerebrovascular disease,
* Respiratory disease,
* Metabolic disease,
* Active inflammatory bowel or renal disease,
* Malignancy,
* Recent steroid treatment (within 6 months) or hormone replacement therapy,
* Clotting dysfunction,
* Musculoskeletal or neurological disorders,
* Family history of early (<55y) death from cardiovascular disease

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 0 - 8 weeks
  Comparison of muscle protein synthesis using D2O in young and older individuals and in response to 8 weeks concentric or eccentric exercise training

SECONDARY OUTCOMES:
Tendon protein synthesis | 0 - 8 weeks
  Comparison of tendon protein synthesis in young and older individuals and in response to 8 weeks concentric or eccentric exercise training

OTHER OUTCOMES:
Muscle function | 0 - 8 weeks
  Muscle strength, force and power in young and older individuals and in response to 8 weeks concentric or eccentric exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Marco V Narici, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Derby, Derbyshire, United Kingdom